CLINICAL TRIAL: NCT01380561
Title: A Metabolite Identification, Mass Balance, and Pharmacokinetic Study of a Single Oral Dose of [14C]-Asimadoline Followed by Twice Daily Oral Dosing of 0.5 mg Asimadoline to Healthy Adult Male Volunteers
Brief Title: A Metabolite Identification, Mass Balance, and PK Study of [14C]-Asimadoline to Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tioga Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ASMP1001
Record Dates: First submitted 2011-06-13; First posted 2011-06-27 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: asimadoline; pharmacokinetic; excretion of 14C-derived radioactivity; metabolite profile; 14C-asimadoline; metabolites; single and multiple oral doses
MeSH Terms: interventions — asimadoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Study (Experimental): asimadoline
  Interventions: Drug: asimadoline

INTERVENTIONS:
Drug: asimadoline — 10mg [14]C labelled asimadoline Day 1 then 7 doses 0.5 mg asimadoline bid beginning on Day 2 and ending on Day 5.
  Other Names: EMD 61 753; EMR 63 320

SUMMARY:
This is an open label, single center, metabolite identification, mass balance, and PK study in healthy male volunteers.

DETAILED DESCRIPTION:
This is an open label, single center, metabolite identification, mass balance, and PK study in healthy male volunteers. The purposes of this study is to determine the excretion of total [14C] derived radioactivity and the metabolite profile after a single oral dose of [14C] asimadoline as well as to identify and quantitate the metabolites of asimadoline in plasma, urine, and feces after single and multiple oral doses of asimadoline.

ELIGIBILITY:
Inclusion Criteria:

* Be informed of the nature of the study and have provided written informed voluntary consent
* Be healthy males, at least 18 years of age or the legal age of consent (whichever is greater) and less than 56 years of age
* Have a body mass index (BMI) >=18.0 and <32.0 kg/m2 and weigh at least 50 kg
* Be in good general health with no clinically relevant abnormalities based on the medical history, physical examination, clinical laboratory evaluations (hematology, clinical chemistry, urinalysis), and 12 lead electrocardiogram (ECG) that, in the opinion of the Investigator, would affect subject safety
* Agree to comply with the study procedures and restrictions.

Exclusion Criteria:

* Any disease or condition that might affect drug absorption, metabolism, or excretion, or clinically significant cardiovascular, hematological, renal, hepatic, pulmonary, endocrine, gastrointestinal, immunological, dermatological, neurological, or psychiatric disease
* Receipt of a radioisotope with an effective half-life of 30 days or more within the previous 12 months
* Receipt of any diagnostic radiation procedures with an effective dose exceeding 1 rem in their lifetime
* Occupational exposure to radiation (e.g., those routinely required to wear a radiation monitoring badge)
* Receipt of any radiation treatments/therapy
* History of constipation or infrequent bowel movements (<=6 bowel movements per week on average)
* Known or suspected hypersensitivity or allergic reaction to asimadoline or similar chemical compounds or any of the components of asimadoline tablets
* Chronic use of any systemic medications (with the exception of vitamins taken at standard supplement doses); use of a drug therapy (including herbal preparations, e.g., St. John's wort) known to induce or inhibit hepatic drug metabolism within 30 days before the first dose of study medication; use of prescription medication within 14 days before administration of study medication or over-the-counter products (including natural products) within 7 days before administration of study medication, except for topical products without systemic absorption, unless approved by the Sponsor
* Have smoked cigarettes or used nicotine-containing products over the last 3 months and not able to abstain from smoking for the duration of the confinement period
* If not sterile, cannot agree to use one of the following approved methods of contraception, from check-in until 3 months following Study Completion/Clinic Discharge: a male condom with spermicide; a sterile sexual partner; use by a female sexual partner of an intrauterine device with spermicide; a female condom with spermicide; contraceptive sponge with spermicide; a cervical cap with spermicide; or oral, implantable, transdermal, or injectable contraceptives with a reliable secondary back-up method
* Current history or evidence of drug or alcohol abuse or a positive screen for substances of abuse or alcohol at screening or admission
* Positive screen for hepatitis B surface antigen (HBsAg), hepatitis C antibody, or human immunodeficiency virus (HIV) antibody
* Receipt of an investigational product or device, or participation in a drug research study within a period of 30 days (or 5 half lives of the drug, whichever is longer) before the first dose of study medication
* Blood loss or blood donation of >550 mL within 90 days or plasma donation >500 mL within 30 days before administration of study drug
* Any food allergy, intolerance, restriction, or special diet that, in the opinion of the Investigator, should preclude the subject's participation in this study

Ages: 18 Years to 56 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Amount of [14C]derived radioactivity in urine and feces after a single oral dose of [14C]asimadoline | up to 1 month
Concentration of metabolites of asimadoline in plasma, urine, and feces after single and multiple oral doses of asimadoline. | up to 1 month

SECONDARY OUTCOMES:
Determination of plasma pharmacokinetics (e.g., Cmax, AUC, tmax, t1/2) of asimadoline and major metabolites | up to 1 month
Number of subjects with adverse events | up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Philip Leese, Principal Investigator — Quintiles Phase 1 Unit
Locations (1):
- Quintiles Phase 1 Unit, Overland Park, Kansas, United States